CLINICAL TRIAL: NCT03778619
Title: Multi-center, Open-label, Phase 1/2a Clinical Trial to Evaluate the Efficacy and Safety of Combination Therapy With MG4101 Plus Rituximab in Patient With Relapsed/Refractory Non-Hodgkin's Lymphoma of B-cell Origin
Brief Title: MG4101 Plus Rituximab Including Lymphodepletion in Patient With r/r NHL B-cell Origin
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG4101-NHL-P1
Record Dates: First submitted 2018-11-07; First posted 2018-12-19 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Relapsed Non Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; fludarabine; fludarabine phosphate; Cyclophosphamide; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): 1. Phase 1
     1. MG4101 (Allogeneic Natural Killer cell): i.v bi-weekly
        * Group 1: 1 x 10^7 cells/㎏
        * Group 2: 3 x 10^7 cells/㎏
        * Group 3: 9 x 10^7 cells/㎏
     2. Interleukin-2 (IL-2): s.c bi-weekly with MG4101 at 1X10^6 IU/m2 per day.
     3. Rituximab: 375mg/m2. i.v. weekly for the first 2 cycles only (8 doses). monthly (3-6 cycle)
     4. Lymphodepletion: Fludarabine 20mg/m2 + Cyclophosphamide 250 mg/m2 i.v. D-3, D-2, D-1 of 1st, 3rd, and 5th cycle
  2. Phase 2a Administration of recommended dosage of MG4101 determined from Phase 1 will be applied in Phase 2a. Dosage regimens for lymphodepletion, IL-2 and Rituximab will be the same as Phase 1.
  Interventions: Drug: Rituximab; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: MG4101(allogeneic Natural Killer cell); Drug: Interleukin-2

INTERVENTIONS:
Drug: Rituximab — weekly administration of Rituximab 375mg/m2 during cycle 1 and 2, monthly administration from cycle 3(up to cycle 6)
  Other Names: Mabthera
Drug: Fludarabine — administration of fludarabine 20mg/m2 for 3 consecutive days starting at 3 days before the 1st, 3rd, and 5th cycle of the first rituximab infusion for that cycle
  Other Names: Fludara
Drug: Cyclophosphamide — administration of fludarabine 250mg/m2 for 3 consecutive days starting at 3 days before the 1st, 3rd, and 5th cycle of the first rituximab infusion for that cycle
  Other Names: Endoxan
Biological: MG4101(allogeneic Natural Killer cell) — administration every fortnight for each cycle, beginning with the 1st dose of rituximab for that cycle.
Drug: Interleukin-2 — 1 x 10^6 IU/m2, together with MG4101
  Other Names: proleukin

SUMMARY:
To determine the efficacy and safety of combined therapy of determined MG4101 dose and Rituximab.

DETAILED DESCRIPTION:
This trial will consist of 3 parts; Phase 1 Maximum Tolerated Dose, Phase 1 extended cohort and Phase 2a.

For Phase 1, those who have a confirmed diagnosis of relapsed/refractory Non-Hodgkin's Lymphoma (NHL) of B-cell Origin of any subtype will be considered eligible for enrolment. Each cycle last approximately 28 days.

Once the dose of MG4101 is determined from Phase 1, Phase 2a will commence whereby two subgroups of patients will be enrolled and will similarly receive up to 6 cycles of treatment with the recommended Phase 2a dose of MG4101. The 2 subgroups are patients with indolent and aggressive NHL of B-cell origin respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory NHL of B-cell origin (mature B cell lymphoma according to WHO)* who are not considered candidates for intensive anti-lymphoma therapy.
2. Patients must have received at least 1 prior systemic treatment including anti-CD20 therapy but have received no more than 4 systemic treatments and have:

   1. Relapse/Progression and is not considered as a candidate for autologous stem-cell transplantation or high-dose immuno-chemotherapy with allogenic antibody transplantation.
   2. Or Relapsed/progressed after high-dose immuno-chemotherapy with autologous stem-cell transplantation.
   3. Or Relapsed/progressed after homoplastic stem-cell transplantation performed at least 12 weeks ago from C1V1.

      * For Phase 1 - Any subtype can be enrolled. For Phase 2a - Only below subtype can be enrolled in each group. I. Indolent B-cell NHL: Follicular Lymphoma, Lymphoplasmacytic Lymphoma, Mantle Cell Lymphoma and Marginal Zone Lymphoma II. Aggressive B-cell NHL: Diffuse Large B-cell Lymphoma De novo and Diffuse Large B-cell Lymphoma transformed
3. According to Positron Emission Tomograph(PET)-CT screening, patients having lesion/nodules ≥1 with major axis longer than 1.5 cm and the boundaries are clearly shown.
4. Eastern Cooperative Oncology Group score 0 or 1
5. 20 years or older. Age limit for Phase 1 is 65 and for Phase 2a 80.
6. Expected lifespan ≥ 3 month
7. Patients signed Informed consent form
8. Earlier documented result that showed that the patient is positive for CD20 via immunophenotyping within 6 months of C1V1
9. Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for clinically non-significant toxicities such as alopecia)
10. Those patients who satisfied with following criteria in blood testing, kidney function test and liver function test:

    1. Absolute neutrophil count: Absolute Neutrophil Count ≥ 1,000/ µL (Growth factor support at least 2 weeks prior to C1V1)
    2. Haemoglobin level ≥ 8g/㎗ (Blood transfusion at least 2 weeks prior to C1V1)
    3. Platelet count ≥75,000/µL (Growth factor support/blood transfusion at least 2 weeks prior to C1V1)
    4. Total bilirubin < 3.0㎎/㎗
    5. Aspartate aminotransferase(AST) or Alanine Aminotransferase(ALT) ≤ 2.5 x upper normal limit (UNL)
    6. Creatinine clearance (as estimated by Cockcroft Gault) ≥ 30 mL/min

Exclusion Criteria:

1. Patients considered appropriate to have stem-cell transplantation after high-dose chemotherapy as salvage therapy.
2. Patient with Central Nervous System(CNS) lymphoma or any involvement of the CNS.
3. Patients who had a prior history of another malignancy over the last 5 years.
4. Patients with impaired organ functions deemed as significant by investigators.
5. Patients who had prior allogeneic Natural Killer cell treatment.
6. Chronic or active infectious diseases required to be treated at the time of Investigational Product administration, including Cytomegalovirus(CMV) prophylactic therapy.
7. Had human immunodeficiency virus (HIV)-positive serology.
8. HBsAg or Hepatitis B virus(HBV) DNA positive or had Hepatitis C virus(HCV) antibodies
9. Patients who received anti-CD20 cancer chemotherapy or immunoglobulin within 4 weeks of C1V1.
10. Patients who received another investigational drug within 4 weeks of C1V1.
11. Patients with acute graft-versus-host disease(GvHD) ≥Grade 3 or extensive chronic GvHD within 2 weeks of C1V1.
12. High-dose stem cell support treatment carried out within 6 months of C1V1.
13. Radioimmunotherapy within 4 weeks of C1V1.
14. Patients with major surgery within 4 weeks of C1V1.
15. Patients required to have treatment as having severe diseases such as severe heart failure or uncontrolled severe heart disease and considered not to be appropriate to participate in this trial by investigator's decision.
16. Patients on enzyme inducing agents.
17. Patients who have a plan to have vaccination during the trial.
18. Patients with sensitivity to Interleukin-2, cyclophosphamide or fludarabine.
19. Patients with urinary outflow obstruction
20. Patients with history of abnormal cardiac or pulmonary function tests in 6 months prior to screening visit (Clinically Significant)
21. Patients with history of solid organ allografts
22. Patients with pre-existing or initial presentation of autoimmune disease or inflammatory disorders, such as Crohn's disease, scleroderma, thyroiditis, inflammatory arthritis, diabetes mellitus, oculo-bulbar myasthenia gravis, crescentic Immunoglobulin A(IgA) glomerulonephritis, cholecystitis, cerebral vasculitis, Stevens-Johnson syndrome and bullous pemphigoid, due to possible exacerbation with IL-2
23. Concomitant treatment with other cardiotoxic inducing agents
24. Patients who are allergic to Rituximab, Rituximab's excipient (sodium citrate, polysorbate 80, sodium chloride, sodium hydroxide, hydrochloric acid) or other proteins same as Rituximab.
25. From the day of participation of this trial to 12 months from the day of final administration of Investigational Product, patients who are unable or unwilling to use appropriate contraceptive methods. (Condom, diaphragm, Intrauterine Device, hormonal oral contraceptive use, or male partner with vasectomy)
26. Pregnant or lactating women. (Breast-feeding cannot be done within 12 months after final Investigational Product administration)
27. Patients suspected to have currently known or suspected alcohol abuse or drug abuse according to investigator's decision.
28. According to investigator's judgement, protocols cannot be followed.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Phase I - Maximum Tolerated Dose of the dose of MG4101 in combination with Rituximab | 28 days
  Dose-Limiting Toxicity assessment
Phase II - Objective Response Rate | up to 3 years
  central review by Positron Emission Tomograph-CT

SECONDARY OUTCOMES:
Phase I - Objective Response Rate | 1 years
  investigator review by Positron Emission Tomograph-CT
Phase II - Complete Response | up to 3 years
  Complete Response Rate
Phase II -Partial Response | up to 3 years
  Partial Response rate
Phase II - Overall Survival | up to 3 years
  every 12 weeks after End Of Treatment
Phase II - Time To Progression | up to 3 years
  every 12 weeks after End Of Treatment
Phase II - Time to Response | up to 3 years
  every 12 weeks after End Of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, Dr., Principal Investigator — Samsung Medical Center
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National Univ. Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No